CLINICAL TRIAL: NCT03313518
Title: Therapeutic Role of Transcranial Direct Current Stimulation (tDCS) in Alzheimer Patients, Double Blind Placebo Controlled Clinical Trial
Brief Title: Therapeutic Role of Transcranial DCS in Alzheimer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman M. Khedr, Clinical Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tDCS in Alzheimer
Record Dates: First submitted 2017-10-14; First posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Alzheimer Disease
Keywords: tDCS, Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anodal tDCS (Active Comparator): Transcranial Direct Current Stimulation using anodal electrode, 15 patients received real anodal tDCS 2mA for 20 minutes for 10 consecutive days.
  Interventions: Device: tDCS
- sham group (Sham Comparator): Fifteen patients received sham anodal tDCS 2mA for 20 minutes for 10 consecutive days.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: tDCS — 15 patients received real anodal tDCS for 20 minutes daily for 10 consecutive days.
  Arms: Anodal tDCS
Device: Sham tDCS — 15 patients received sham anodal tDCS for 20 minutes daily for 10 consecutive days.
  Arms: sham group

SUMMARY:
The aim of this study is to evaluate the oxidative stress and brain damage biomarkers induced by tDCS in patients with AD and to assess the long term neurophysiological and behavioral effects after repeated daily tDCS sessions for 10 days. Thirty AD patients diagnosed according to 2011 McKhann criteria will be randomly assigned to receive 10 real anodal tDCS or sham at 2mA intensity for 20 minutes per session daily. All patients will be evaluated at baseline, at the end of the sessions and 1, 2, and 3 months later with neurophysiological and behavioral examination.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the oxidative stress and brain damage biomarkers induced by tDCS in patients with AD and to assess the long term neurophysiological and behavioral effects after repeated daily tDCS sessions for 10 days. Thirty AD patients diagnosed according to 2011 McKhann criteria will be randomly assigned to receive 10 real anodal tDCS or sham at 2mA intensity for 20 minutes per session daily. Patients were classified into two groups using closed envelope. One group will receive 10 sessions real tdcs and other group will receive sham tdcs.

The study will be a double-blind, placebo controlled, within subject, parallel design.

tDCS will be delivered bilaterally by a constant current electrical stimulator connected to a pair of sponge electrodes. The investigators will use a non-cephalic reference electrode for tDCS: stimulating electrode will be placed over the left temporo-parietal lobe for 20 minutes and then over the right temporoparietal lobe for another 20 minutes in AD patients, while the reference electrode will be placed over the right deltoid muscle. The stimulating current will be anodal DC at 2 mA intensity delivered for 20 minutes per session for 10 days. All patients will be evaluated at baseline, at the end of the treatment and 1 and 2,and 3months later with neuropsychological and behavioural examination.

ELIGIBILITY:
Inclusion Criteria:

* All subject were diagnosed with Probable AD according to NINCDS/ADRDA Criteria for Alzheimer's Disease.
* Onset age > 60.
* All 4 grandparents are of Ashkenazi Jewish origin as declared by the subject.
* Subject or subject's legal representative has signed the informed consent form.

Exclusion Criteria:

* All subjects who were diagnosed with Possible AD according to NINCDS/ADRDA Criteria for Alzheimer's Disease.
* Subjects who were diagnosed with dementia due to other diseases, or with AD and contribution of other disorders (Mixed dementia):
* Brain CT/MRI suggesting alternative diagnoses, such as intracranial space occupying lesions, vascular lesion of the brain, white matter lesion, or hydrocephalus.
* Subjects who had known carrier of a blood transmitted infectious disease or suffers from conditions in which phlebotomy is contra-indicated.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-08-12 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
Change in measurement of improvement in cognitive function by using MMSE | three months
  Change in measurement of improvement in cognitive function by using MMSE
Change in measurement of improvement in cognitive function by cornell Scale | Three months
  Change in measurement of improvement in cognitive function by cornell Scale

SECONDARY OUTCOMES:
The change of measurement of brain damage biomarkers modulation in plasma (i.e. Tau, Beta-Amyloid, Lipid Peroxidation) cornell Scale | ten days
  measure the change of brain damage biomarkers modulation in plasma (i.e. Tau, Beta-Amyloid, Lipid Peroxidation)

CONTACTS AND LOCATIONS:
Overall Officials: Eman M. Khedr, MD, Principal Investigator — Professor of Neurology, Faculty of Medicine, Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khedr EM, Salama RH, Abdel Hameed M, Abo Elfetoh N, Seif P. Therapeutic Role of Transcranial Direct Current Stimulation in Alzheimer Disease Patients: Double-Blind, Placebo-Controlled Clinical Trial. Neurorehabil Neural Repair. 2019 May;33(5):384-394. doi: 10.1177/1545968319840285. Epub 2019 Apr 3. PMID 30940012